CLINICAL TRIAL: NCT04604717
Title: Effect of Exercise Training on Salivary Immunoglobulin A in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Austin Health (Other Government); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110314; IBAS110314 (Other Grant/Funding Number: IBAS13)
Record Dates: First submitted 2014-03-11; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: COPD
Keywords: COPD,; Pulmonary rehabilitation,; Airway immunity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary rehabilitation (Experimental): 8 weeks of pulmonary rehabilitation (twice weekly training) Exercise and education sessions accompanied by home exercise program
  Interventions: Other: Pulmonary rehabilitation
- Control group (No Intervention): Usual medical treatment for 8 week period

INTERVENTIONS:
Other: Pulmonary rehabilitation — 8 weeks of exercise training (twice weekly) of education and exercise
  Arms: Pulmonary rehabilitation

SUMMARY:
The purpose of this study is to determine whether whole body exercise training alters the immunity in the lungs of people with COPD and reduces the incidence of chest infections over the longer term.

DETAILED DESCRIPTION:
Patients will undertake an 8 weeks pulmonary rehabilitation program of exercise and education. Those who decline to take part in pulmonary rehabilitation will have the same outcome measures collected at the same timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (FEV1/FVC < 70), smoking Hx of minimum of 10 pack years

Exclusion Criteria:

* Diagnosis of asthma, bronchiectasis, attendance at pulmonary rehabilitation within last 12 months, exacerbation of COPD within last 4 weeks

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Salivary Immunoglobulin A levels | Change over 8 weeks
  SIgA

SECONDARY OUTCOMES:
Change in circulatory inflammatory markers | Change over 8 weeks
Change in physical activity levels | Change over 8 weeks
Health status | Change over 8 weeks
  COPD assessment test
Exercise capacity (6MWT) | Change over 8 weeks
  Distance walked in 6 minutes
Number of acute exacerbations | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Holland, PhD, Principal Investigator — Alfred Health, La Trobe University
Locations (2):
- Australia (2):
  - Alfred Health, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria